CLINICAL TRIAL: NCT06324747
Title: Soft Tissue Stability in Immediate Implant Placement Using the Vestibular Socket Therapy Versus Conventional Flap in Type II Extraction Sockets in the Esthetic Zone: A Randomized Clinical Trial
Brief Title: Soft Tissue Stability in Immediate Implant Placement Using (VST) Versus Conventional Flap in Type II Extraction Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Mohamed shawky, Dentist (BDS), British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-046
Record Dates: First submitted 2023-12-04; First posted 2024-03-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Badly Broken Tooth in a Socket Type II Eligible to be Replaced by Immediate Implant

STUDY DESIGN:
Intervention Model Description: Two equal parallel groups with a 1:1 allocation ratio to receive either vestibular socket therapy (test group) or to be treated with conventional mucoperiosteal flap (control group).
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the differences in techniques, the operating surgeon can not be blinded to the procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other): Control group will have a full thickness flap, followed by an immediate implant placement using a surgical guide. Then a guided bone regeneration will be achieved by bone graft (autogenous bone chips and xenograft particles and a membrane barrier 1 mm thickness will be applied. The membrane shield then will be stabilized to the apical bone using 2 membrane tacks, customized healing abutment will be connected , then, the elevated flap will be sutured to its original position.
  Interventions: Procedure: conventional full thickness flap
- Test group (Active Comparator): Elaskary Vestibular socket therapy instruments will be used for the intervention, A 1 cm long vestibular access incision at the allocated hopeless tooth will be made at the base of the hopeless tooth to the adjacent teeth. The vestibular pouch will then be dissected in an incisal direction exposing the total socket area and allowing direct access to the socket environment. An immediate implant will be installed using a surgical guide. A membrane shield 1 mm thick will be, trimmed, and tucked through the vestibular access incision starting at 1 mm beyond the socket orifice and reaching to the apical area of the socket. The gap and/ or the defect between the implant body and the shield will then be filled with the same grafting components so the control group. Finally, the vestibular incision will be secured with sutures. The socket will be sealed with a customized healing abutment.
  Interventions: Procedure: Vestibular socket therapy

INTERVENTIONS:
Procedure: Vestibular socket therapy — Vestibular socket therapy will be used for the intervention.
  Other Names: VST
  Arms: Test group
Procedure: conventional full thickness flap — reflecting the mucoperiosteum to access the extraction socket
  Arms: Control group

SUMMARY:
This study compare between the vestibular socket therapy (VST) and the traditional mucoperiosteal flap reflection in immediate implant placement in type II extraction socket in the esthetic zone.

The technique of vestibular socket therapy (VST), introduced by Elaskry, enables the placement of implants immediately while simultaneously rehabilitating the entire socket, resulting in excellent esthetic and functional outcomes that meet the expectations of patients. VST involves socket augmentation through a minimally invasive vestibular access incision, eliminating the need for the traditional mucoperiosteal flap reflection, regardless of the extent of socket compromise.

DETAILED DESCRIPTION:
Several methods have been suggested for the treatment of class 2 socket types with immediate implant placement. One such technique is the immediate dento-alveolar restoration (IDR), which involves the incorporation of a tuberosity bone graft into the buccal defect, restoring the missing buccal bone walls. However, this technique has some limitations, including the lack of graft stabilization to the host bed, the high rate of bone graft remodeling, and the limited availability of tuberosity bone when wisdom teeth are present.

In contrast, Buser D. extensively researched the early implant placement method. This approach involves extracting the tooth and then waiting for a delay period of 8-12 weeks. According to the authors, this timeframe allows for the development of ample keratinized tissues, the elimination of socket infection, and the occurrence of post-extraction bone remodeling.

In contrast, both early placement and contour augmentation procedures have demonstrated certain drawbacks. These include the collapse of socket walls in both horizontal and vertical directions after tooth extraction, the need for a lengthy treatment duration that can extend up to 8 months, the challenges of maintaining provisional restorations during this extended period, and the potential for post-restorative socket tissue recession due to the reflection of the mucoperiosteal flap . As a result, achieving a successful esthetic treatment outcome becomes difficult to predict.

The technique of vestibular socket therapy (VST), introduced by Elaskry et al. , enables the placement of implants immediately while simultaneously rehabilitating the entire socket, resulting in excellent esthetic and functional outcomes that meet the expectations of patients. VST involves socket augmentation through a minimally invasive vestibular access incision, eliminating the need for the traditional mucoperiosteal flap reflection, regardless of the extent of socket compromise .

The procedure involves making a horizontal incision in the vestibule at the base of the mucogingival junction of the extracted tooth. This is followed by implant placement without the need for a flap, grafting the compromised socket walls through the vestibular access incision. The labial bone defect, which has been grafted with a bone graft, is then protected using a cortical equine membrane, and finally, the socket opening is sealed with a customized healing collar.

ELIGIBILITY:
Inclusion Criteria:

* Hopeless maxillary tooth in the esthetic region missing coronal tooth structure
* Type II socket (deficient labial plate of bone and intact overlying soft tissues)
* Adequate palatal bone, ≥ 3 mm apical bone to engage the immediately placed implants

Exclusion Criteria:

* Smokers
* Pregnant women
* Patients with systemic diseases
* History of chemotherapy or radiotherapy within the past 2 years.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Soft Tissue Stability | 8 months
  it will be measured digitally using the intraoral scanner. A preoperative scanning, immediate postoperative, 2 months postoperative and 8 months postoperative scanning will be done.
  Tool to be used: 3shape trios 4
  what will be assessed:
  * gingival recession
  * loss of interdental papillae height
  Data will be measured in millimeters

SECONDARY OUTCOMES:
Bone Regeneration | 8 months
  measuring the thickness of the labial plate of bone.
  It will be measured preoperatively, immediate postoperative to measure the amount of the augmented bone, 2 months postoperatively and 8 months post operative.
  Tool to be used: cone beam computed tomography (cbct)

OTHER OUTCOMES:
Pink Esthetic Score (PES) | 8 months
  The PES is based on seven variables: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deﬁciency, soft tissue color and soft tissue texture. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shawky, BDS, Principal Investigator — The British University in Egypt
Locations (1):
- The British university in Egypt, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP